CLINICAL TRIAL: NCT00928395
Title: Sustained Therapeutic Effects of Percutaneous Tibial Nerve Stimulation
Brief Title: Modified Extension Study to the SUmiT Trial: Evaluation of Long Term Therapy With Percutaneous Tibial Nerve Stimulation (PTNS) for Overactive Bladder Symptoms
Acronym: STEP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Uroplasty, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPC121908
Record Dates: First submitted 2009-06-24; First posted 2009-06-26 (Estimated); Results first posted 2013-05-16 (Estimated); Last update posted 2013-05-16 (Estimated); Status verified 2013-04

CONDITIONS: Urinary Bladder, Overactive
Keywords: Urgent PC; Overactive Bladder; SUmiT Trial; Overactive Urinary Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive

ARMS (1):
- Urgent PC (Active Comparator): The Urgent PC Neuromodulation System is a minimally invasive neuromodulation system designed to deliver retrograde access to the sacral nerve through percutaneous electrical stimulation of the tibial nerve. The method of treatment is referred to as Percutaneous Tibial Nerve Stimulation (PTNS).
  Interventions: Device: Urgent PC

INTERVENTIONS:
Device: Urgent PC — The Urgent PC Neuromodulation System is a minimally invasive neuromodulation system designed to deliver retrograde access to the sacral nerve through percutaneous electrical stimulation of the tibial nerve. The method of treatment is referred to as Percutaneous Tibial Nerve Stimulation (PTNS).

SUMMARY:
This is a modified extension study to the SUmiT protocol UPC082008 (NCT00534521) to observe and evaluate long term therapy with PTNS on overactive bladder symptoms. Subjects must have completed the 12 weekly treatments of the original protocol, the 13 week follow up assessment, be randomized to the PTNS arm, and be considered a positive responder with moderate or marked improvement in the SUmiT Trial to be enrolled in this study. All consenting responders will continue with active PTNS therapy at an initially prescribed protocol for approximately 3 months followed by individualized symptom-based frequency of visits as determined by the subject along with their treating clinician, for up to a total of 33 months post initial 12-week therapy for a total of 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who signed the informed consent and were eligible to participate in the original SUmiT Trial
* Subjects who were randomized and treated with the active PTNS therapy during their participation in the original SUmiT Trial
* Subject must be a positive responder from initial 12 weekly treatments as prescribed in original SUmiT Trial - 13 week GRA questionnaire must indicate "moderately" or "markedly improved" on question #1 of GRA
* Subjects must not have started any antimuscarinics treatment since completion of original SUmiT Trial
* Subjects must not have started any urologic Botox treatment since completion of original SUmiT Trial
* Subjects must remain off all antimuscarinics throughout participation in trial
* Subjects must initiate PTNS maintenance therapy within 2 weeks of their last PTNS treatment as part of SUmiT protocol UPC082008
* Capable of giving informed consent
* Capable and willing to follow all study-related procedures for up to 33 months for a total participation of 3 years

Exclusion Criteria:

* Pregnant as confirmed by urine pregnancy test, or plans to become pregnant during the study period
* Subjects who were not able or willing to follow original SUmiT Trial study schedule

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-01; Primary Completion 2012-09 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Peters, MD, Principal Investigator — Beaumont Hospital
Locations (12):
- United States (12):
  - Gregory L. Davis, M.D., FACOG, Inc., Chico, California
  - Greenwich Urological Associates, P.C., Greenwich, Connecticut
  - Specialists in Urology, Naples, Florida
  - Grand Rapids Women's Health DBA Female Pelvic Medicine & Urogynecology Institue of Michigan, Grand Rapids, Michigan
  - Mercy Health Partners at the Lakes, Muskegon, Michigan
  - Beaumont Hospital, Royal Oak, Michigan
  - Urology Health Center, PC, Fremont, Nebraska
  - Capital Region Urological Surgeons, PLLC, Albany, New York
  - Central Missouri Women's Healthcare, LLC, White Plains, New York
  - Alliance Urology Specialists, Greensboro, North Carolina
  - Virginia Urology, Richmond, Virginia
  - Athena Urology, Issaquah, Washington

REFERENCES:
- [Derived] Peters KM, Carrico DJ, MacDiarmid SA, Wooldridge LS, Khan AU, McCoy CE, Franco N, Bennett JB. Sustained therapeutic effects of percutaneous tibial nerve stimulation: 24-month results of the STEP study. Neurourol Urodyn. 2013 Jan;32(1):24-9. doi: 10.1002/nau.22266. Epub 2012 Jun 5. PMID 22674493

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited by investigator sites.
Period: Overall Study
Arm/Group | Urgent PC
Started | 50
Completed | 29
Not Completed | 21

BASELINE CHARACTERISTICS:
Arm/Group | Urgent PC
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 26
  >=65 years | 24
Age Continuous [Mean (Standard Deviation); unit: years] | 60.5 (15.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39
  Male | 11
Region of Enrollment [Number; unit: participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Reporting "Moderately" or "Markedly" Improved on the Global Response Assessment (GRA) at 36 Months as Compared to Baseline
Description: The GRA asked patients, "Compared to the last time you completed this questionnaire, how would you rate your bladder symptoms now?" and was a 7-level Assessment (markedly improved, moderately improved, slightly improved, no change, slightly worse, moderately worse, markedly worse).
Time Frame: 36 months total
Measure: Number (95% Confidence Interval); unit: Proportion of Patients
Arm/Group | Urgent PC
Number analyzed (Participants) | 50
Proportion of Patients | .77 [.64 to .90]

2. Secondary Outcome: GRA Subset of Individual Bladder Symptom Components to Include Urgency, Frequency and Urge Incontinence.
Time Frame: every three months for 36 months
Reporting Status: Not Posted

3. Secondary Outcome: Change in OAB-q and SF-36 Questionnaires.
Time Frame: every three months for 36 months
Reporting Status: Not Posted

4. Secondary Outcome: Change in Voiding Diary Parameters.
Time Frame: every three months for 36 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Urgent PC
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 1/50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Urgent PC (N=50)
Bleeding at needle site (Surgical and medical procedures) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No